CLINICAL TRIAL: NCT00737074
Title: Macular Hole in Proliferative Diabetic Retinopathy With Fibrovascular Proliferation
Brief Title: Macular Hole in Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chung-May Yang/Department of Opthalmology, National Taiwan University Hospital, Department of Opthalmology, National Taiwan University Hospital
Other Study IDs: 200806056R
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Macular Hole; Proliferative Diabetic Retinopathy
Keywords: Fibrovascular proliferation; Internal limiting membrane peeling; Macular detachment; Macular hole; Proliferative diabetic retinopathy.
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Macular hole in proliferative diabetic retinopathy with fibrovascular proliferation may have unique features. Internal limiting membrane peeling facilitates hole closure only in cases with shallow macular detachment. Final vision is associated with preoperative visual acuity and degree of macula elevation.

DETAILED DESCRIPTION:
From January 2002 to December 2007 consecutive patients undergo pars plana vitrectomy for diabetic fibrovascular proliferation and the medical and surgical records are reviewed.

Diabetic fibrovascular proliferation associated with macular hole that had undergone pars plana vitrectomy with a minimum of 6 months of post-operative follow-up will be retrospectively reviewed. Cases fulfilling the indication criteria will be selected for the study All operations had been performed following the same principle and techniques.

Demographics and clinical findings of each case will be recorded including age, sex, involved eye, duration of macular hole, intraoperative diagnosis, extent of vitreo-retinal adhesion and detachment, morphology of macular hole, and relationship of macular hole to posterior hyaloid and fibrovascular proliferation. Data regarding treatment of macular hole, final opening or closure of macular hole, and duration of postoperative follow-up will also be compiled. Results of ophthalmological examinations, including pre- and post-operation best corrected visual acuity, intraocular pressure, and intravitreal tamponade material will be recorded. Optical coherence tomography (OCT) findings will be categorized and recorded. Retinal detachment severity will be classified as: no traction retinal detachment (TRD) or TRD within arcade (grade 1); TRD outside arcade, but not to or beyond the equator (grade 2); and RD extended to the periphery in at least 1 quadrant (grade 3). The degree of macular elevation surrounding the macular hole will be classified into three grades according to pre- or intra-operative observation: shallow: barely visible macular detachment with or without fine retinal folds and with underlying choroidal patterns still identifiable through the detached retina; moderate: obvious detachment with folds and loss of visualization of underlying choroidal patterns; and high: convex shaped or dome shaped detachment with wavy configuration in the macular area. Extent of fibrovascular proliferation will be separated into 3 grades: grade 1: focal adhesions only; grade 2: broad adhesion at more than 1 site or vitreous-retinal adhesion at disc, macula or arcade; and grade 3: vitreous-retinal attachment extending to the periphery.

Statistical Analysis To examine the significance of various clinical findings in relation to final macular hole closure rate, statistical analysis of the data is performed with chi-squared test or Fisher's exact test. To further verify the clinical characteristics and treatments that affecting macular hole closure, multivariate logistic regression analysis is performed to determine the significance of the following factors: age, sex, operation eye, duration of macular hole, RD extent, submacular fluid level, extent of fibrovascular proliferation, macular hole shape, and intravitreal tamponade materials. An association of post-operative best-corrected visual acuity with other study variables is assessed by multiple lineal regression analysis, using backward Wald's criteria, taking post-operation best-correted visual acuity as the dependent variable. All of the statistical analyses are performed using STATA 8.2 software (StataCorp LP, College Station, Texas, USA). A P value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* From January 2002 to December 2007 consecutive patients undergo pars plana vitrectomy for diabetic fibrovascular proliferation and the medical and surgical records are reviewed.
* Indications for surgery had been the severe complications of diabetic retinopathy and not the mere presence of macular hole alone.
* Macular hole is found either preoperatively or during operation.
* All cases are included in the study have attached retina postoperatively.

Exclusion Criteria:

* Cases with recurrent rhegmatogenous detachment or post-operative dense cataract without lens extraction.
* Follow-up duration of patients less than 3 months .
* Incomplete medical records.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paitient with proliferative diabetic retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2002-01; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Final opening or closure of macular hole | Six months

SECONDARY OUTCOMES:
Post-operation best corrected visual acuity | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Chung-May Yang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Ophthalmology, National Taiwan University Hospital, Taipei, Taiwan